CLINICAL TRIAL: NCT05381350
Title: A Randomized, Double-blind, Active-controlled Clinical Trial, as Well as an Immuno-bridging Clinical Trial by Parallel Testing Previous Serum After Primary Immunization, to Evaluate the Immunogenicity and Safety of Booster Immunization of COVID-19 Vaccine (Vero Cell), Inactivated (Omicron Variant) in Healthy People Aged 18 Years and Above
Brief Title: Immunogenicity and Safety of Booster Immunization of COVID-19 Vaccine (Vero Cell), Inactivated (Omicron Variant) in Healthy People Aged 18 Years and Above
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sinovac Research and Development Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sinovac Biotech Co., Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PRO-onCOV-3001
Record Dates: First submitted 2022-05-18; First posted 2022-05-19 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Vaccines; sinovac COVID-19 vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Experimental group aged 18-59 years and received 2 doses of COVID-19 vaccine（CZ strain） (Experimental): 400 participants aged 18-59 years and received 2 doses of COVID-19 vaccine（CZ strain） will receive one dose of inactivated COVID-19 vaccine (Omicron variant).
  Interventions: Biological: COVID-19 Vaccine (Vero cell), Inactivated (Omicron variant)
- Control Group aged 18-59 years and received 2 doses of COVID-19 vaccine（CZ strain） (Active Comparator): 200 participants aged 18-59 years and received 2 doses of COVID-19 vaccine（CZ strain） will receive one dose of inactivated COVID-19 vaccine（CZ strain）.
  Interventions: Biological: COVID-19 Vaccine (Vero cell), Inactivated (CZ strain)
- Experimental group aged 60 years and above and received 2 doses of COVID-19 vaccine（CZ strain） (Experimental): 100 participants aged 60 years and above and received 2 doses of COVID-19 vaccine（CZ strain） will receive one dose of inactivated COVID-19 vaccine (Omicron variant).
  Interventions: Biological: COVID-19 Vaccine (Vero cell), Inactivated (Omicron variant)
- Control Group aged 60 years and above and received 2 doses of COVID-19 vaccine（CZ strain） (Active Comparator): 50 participants aged 60 years and above and received 2 doses of COVID-19 vaccine（CZ strain） will receive one dose of inactivated COVID-19 vaccine（CZ strain）.
  Interventions: Biological: COVID-19 Vaccine (Vero cell), Inactivated (CZ strain)
- Experimental group aged 18-59 years and received 3 doses of COVID-19 vaccine（CZ strain） (Experimental): 400 participants aged 18-59 years and received 3 doses of COVID-19 vaccine（CZ strain） will receive one dose of inactivated COVID-19 vaccine (Omicron variant).
  Interventions: Biological: COVID-19 Vaccine (Vero cell), Inactivated (Omicron variant)
- Control Group aged 18-59 years and received 3 doses of COVID-19 vaccine（CZ strain） (Active Comparator): 200 participants aged 18-59 years and received 3 doses of COVID-19 vaccine（CZ strain） will receive one dose of inactivated COVID-19 vaccine（CZ strain）.
  Interventions: Biological: COVID-19 Vaccine (Vero cell), Inactivated (CZ strain)
- Experimental group aged 60 years and above and received 3 doses of COVID-19 vaccine（CZ strain） (Experimental): 100 participants aged 60 years and above and received 3 doses of COVID-19 vaccine（CZ strain） will receive one dose of inactivated COVID-19 vaccine (Omicron variant).
  Interventions: Biological: COVID-19 Vaccine (Vero cell), Inactivated (Omicron variant)
- Control Group aged 60 years and above and received 3 doses of COVID-19 vaccine（CZ strain） (Active Comparator): 50 participants aged 60 years and above and received 3 doses of COVID-19 vaccine（CZ strain） will receive one dose of inactivated COVID-19 vaccine（CZ strain）.
  Interventions: Biological: COVID-19 Vaccine (Vero cell), Inactivated (CZ strain)
- Historical control group (Active Comparator): Backup serum samples will be selected from 250 healthy adult subjects aged 26-45 years who received two doses of inactivated COVID-19 vaccine(CZ strain)from clinical trial of lot-to-lot consistency of an inactivated SARS-CoV-2 Vaccine(Pro-NCOV-4001) to detect neutralizing antibodies against the CZ, Delta and Omicron strains.
  Interventions: Biological: COVID-19 Vaccine (Vero cell), Inactivated (CZ strain)

INTERVENTIONS:
Biological: COVID-19 Vaccine (Vero cell), Inactivated (Omicron variant) — The COVID-19 Vaccine (Vero cell), Inactivated (Omicron variant)was manufactured by Sinovac Research& Development Co., Ltd.1200SOU inactivated SARS-CoV-2 Omicron strain in 0.5ml of aluminium hydroxide solution per injection.
  Arms: Experimental group aged 18-59 years and received 2 doses of COVID-19 vaccine（CZ strain）; Experimental group aged 18-59 years and received 3 doses of COVID-19 vaccine（CZ strain）; Experimental group aged 60 years and above and received 2 doses of COVID-19 vaccine（CZ strain）; Experimental group aged 60 years and above and received 3 doses of COVID-19 vaccine（CZ strain）
Biological: COVID-19 Vaccine (Vero cell), Inactivated (CZ strain) — The COVID-19 vaccine,inactivated was manufactured by Sinovac Research& Development Co., Ltd.600SU inactivated SARS-CoV-2 CZ strain virus in 0.5 mL of aluminium hydroxide solution per injection.
  Other Names: CoronaVac
  Arms: Control Group aged 18-59 years and received 2 doses of COVID-19 vaccine（CZ strain）; Control Group aged 18-59 years and received 3 doses of COVID-19 vaccine（CZ strain）; Control Group aged 60 years and above and received 2 doses of COVID-19 vaccine（CZ strain）; Control Group aged 60 years and above and received 3 doses of COVID-19 vaccine（CZ strain）; Historical control group

SUMMARY:
This is a randomized, double-blind, active-controlled Phase Ⅲ clinical trial, as well as an immuno-bridging clinical trial by parallel testing previous serum after primary immunization of COVID-19 vaccine (Vero cell), inactivated (Omicron variant). The main purpose of this study is to evaluate the superiority of immunogenicity against SARS-CoV-2 Omicron strain induced by one-dose booster immunization of inactivated COVID-19 vaccine (Omicron variant), developed by Sinovac Research and Development Co., Ltd.in subjects who have received two- or three-dose Prototype COVID-19 vaccine （CZ strain）, compared with one-dose booster of Prototype COVID-19 vaccine （CZ strain） in subjects who have received three-dose Prototype COVID-19 vaccine （CZ strain）, and to evaluate the non-inferiority of immunogenicity against SARS-CoV-2 Omicron strain induced by one-dose booster immunization of inactivated COVID-19 vaccine (Omicron variant), developed by Sinovac Research and Development Co., Ltd., in subjects who have received two- or three-dose Prototype COVID-19 vaccine, compared with the immunogenicity against SARS-CoV-2 Prototype strain induced by two-dose Prototype COVID-19 vaccine（CZ strain）after primary immunization.

DETAILED DESCRIPTION:
This study is a single-center, randomized, double-blind, active-controlled Phase Ⅲ clinical trial, as well as an immuno-bridging clinical trial by parallel testing previous serum after primary immunization of COVID-19 vaccine (Vero cell), inactivated (Omicron variant). The main purpose of this study is to evaluate the superiority of immunogenicity against SARS-CoV-2 Omicron strain induced by one-dose booster immunization of inactivated COVID-19 vaccine (Omicron variant)developed by Sinovac Life Sciences Co., Ltd.in subjects who have received two- or three-dose COVID-19 vaccine（CZ strain）, compared with one-dose booster of COVID-19 vaccine（CZ strain）in subjects who have received three-dose COVID-19 vaccine（CZ strain）and to evaluate the non-inferiority of immunogenicity against SARS-CoV-2 Omicron strain induced by one-dose booster immunization of inactivated COVID-19 vaccine (Omicron variant), developed by Sinovac Life Sciences Co., Ltd, in subjects who have received two- or three-dose COVID-19 vaccine（CZ strain）,compared with the immunogenicity against SARS-CoV-2（CZ strain）induced by two-dose COVID-19 vaccine（CZ strain）primary immunization. This clinical trial consists of two stages. A total of 1750 healthy subjects will be enrolled including 1500 healthy subjects aged 18 years and older who have received 2 or 3 doses of the COVID-19 vaccine（CZ strain）（750 population were vaccinated with 2 doses and 3 doses of COVID-19 vaccine（CZ strain）respectively）in stage I of the clinical trial,250 subjects in stage Ⅱ of the clinical trial.

Stage I of the clinical trial:1500 healthy subjects （750 population were vaccinated with 2 doses or 3 doses of COVID-19 vaccine（CZ strain）respectively）who have received two or three doses of the prototype (CZ strain) COVID-19 vaccine, including 1200 subjects aged 18~59 years old and 300 subjects aged 60 years and above. Subjects in each age group will be randomly divided into experimental group and control group in a ratio of 2:1. Subjects in the experimental group will receive one dose of inactivated COVID-19 vaccine (Omicron variant), and subjects in the control group will receive one dose of COVID-19 vaccine（CZ strain）.

Stage Ⅱ of the clinical trial:Backup serum samples will be selected from 250 healthy adult subjects aged 26-45 years who received two doses of inactivated COVID-19 vaccine(CZ strain)from clinical trial of lot-to-lot consistency of an inactivated SARS-CoV-2 Vaccine(Pro-NCOV-4001).

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18 years and above;
* Subjects completed two doses of the prototype COVID-19 vaccine (CZ strain)(the interval between the first dose and the second dose was 1-2 months)or completed 3 doses of prototype COVID-19 vaccine (CZ strain)over 6 months (the interval between the first dose and the second dose was 1-2 months, and the interval between the second dose and the third dose was 6 months or more);
* The subjects can understand and voluntarily sign the informed consent form;
* Provide legal identification and vaccination certificate of prototype COVID-19 vaccine (CZ strain).

Exclusion Criteria:

* History of SARS-CoV-2 infection(laboratory confirmed);
* Close contact with a confirmed COVID-19 (nucleic acid test or antigen test positive patients)within 14 days prior to randomization;
* Received other COVID-19 vaccine in the past except for two or three doses of prototype vaccine;
* Allergy to vaccines or vaccine/placebo ingredients, and serious adverse reactions to vaccines, such as urticaria, dyspnea, angioneuroedema;
* Autoimmune disease and/or blood disease history (including but not limited to systemic lupus erythematosus, thyroidectomy, autoimmune thyroid disease, any form of malignancy, absence of spleen, functional absence of spleen, or splenectomy for any condition),patients with well-controlled type 1 diabetes can be enrolled;
* Serious chronic diseases, such as serious cardiovascular diseases, hypertension, diabetes, liver and kidney diseases, malignant tumors, etc;
* Severe neurological disease (epilepsy, convulsions or convulsions) or mental illness;
* Diagnosed abnormal blood coagulation function (eg, lack of blood coagulation factors, blood coagulopathy, abnormal platelets) or obvious bruising or blood coagulation;
* Immunosuppressive therapy, cytotoxic therapy, inhaled corticosteroids (excluding allergic rhinitis corticosteroid spray therapy, acute noncomplicated dermatitis superficial corticosteroid therapy) in the past 6 months;
* Long-term history of alcohol or drug abuse;
* Received blood products within 3 months prior to receiving the investigational vaccine, or planning to receive the above treatments during the study period;
* Receipt of other investigational drugs in the past 30 days;
* Receipt of attenuated live vaccines in the past 14 days;
* Receipt of inactivated or subunit vaccines in the past 7 days;
* Onset of various acute or chronic diseases within 7 days prior to the study;
* In case of fever on the day of planned trial vaccine inoculation,axillary temperature >37.0°C;
* Women who are breastfeeding, pregnant, or planning to become pregnant during the study period (based on subjects' self-reported and urine pregnancy test results);
* Participating in or planning to participate in clinical trials of other vaccines or drugs;
* According to the investigator's judgment, the subject has any other factors that are not suitable for participating in the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1750 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-09-26 (Actual); Study Completion 2023-03-09 (Actual)

PRIMARY OUTCOMES:
Geometric mean titres (GMTs) and seroconversion rates of the neutralizing antibody to SARS-CoV-2 Omicron strain (BA.1) | 28 days (Day 28) after booster vaccination
  Geometric mean titres (GMTs) and seroconversion rates of the neutralizing antibody to SARS-CoV-2 Omicron strain (BA.1), induced by a booster dose of COVID-19 vaccine (Omicron variant), 28 days (Day 28) after booster vaccination among subjects with two- or three-dose COVID-19 vaccine（CZ strain） ≥6 months before
GMTs and seroconversion rates of the neutralizing antibody to SARS-CoV-2 Omicron strain (BA.1) | 28 days (Day 28) after booster vaccination
  GMTs and seroconversion rates of the neutralizing antibody to SARS-CoV-2 Omicron strain (BA.1), induced by a booster dose of Prototype COVID-19 vaccine, 28 days (Day 28) after booster vaccination among subjects with three-dose Prototype COVID-19 vaccine≥6 months before
GMTs of the neutralizing antibody to SARS-CoV-2 Prototype strain(CZ strain) | 28 days after vaccination of two doses of Prototype COVID-19 vaccine
  GMTs of the neutralizing antibody to SARS-CoV-2 Prototype strain induced by two doses of Prototype COVID-19 vaccine, 28 days after vaccination in previous clinical trial serums

SECONDARY OUTCOMES:
Geometric mean increases (GMIs) and seropositive rates of the neutralizing antibody to SARS-CoV-2 Omicron strain (BA.1), as well as GMTs, GMIs, seroconversion rates and seropositive rates of the neutralizing antibody to SARS-CoV-2 Omicron strain (BA.2) | 28 days (Day 28) after booster vaccination
  Geometric mean increases (GMIs) and seropositive rates of the neutralizing antibody to SARS-CoV-2 Omicron strain (BA.1), as well as GMTs, GMIs, seroconversion rates and seropositive rates of the neutralizing antibody to SARS-CoV-2 Omicron strain (BA.2), induced by a booster dose of COVID-19 vaccine (Omicron variant), 28 days (Day 28) after booster vaccination among subjects with two-dose Prototype COVID-19 vaccine ≥6 months before
GMIs,seroconversion rates seropositive rates of the neutralizing antibody to SARS-CoV-2 Omicron strain (BA.1), as well as GMTs, GMIs, seroconversion rates and seropositive rates of the neutralizing antibody to SARS-CoV-2 Omicron strain (BA.2) | 28 days (Day 28) after booster vaccination
  GMIs and seropositive rates of the neutralizing antibody to SARS-CoV-2 Omicron strain (BA.1), as well as GMTs, GMIs, seroconversion rates and seropositive rates of the neutralizing antibody to SARS-CoV-2 Omicron strain (BA.2), induced by a booster dose of COVID-19 vaccine (Omicron variant) or prototype COVID-19 vaccine, 28 days (Day 28) after booster vaccination among subjects with three-dose Prototype COVID-19 vaccine ≥6 months before
GMTs, GMIs, seroconversion rates and seropositive rates of the neutralizing antibody to SARS-CoV-2 Omicron strain (BA.1, BA.2), Prototype strain and Delta strain | 28 days (Day 28) after booster vaccination
  GMTs, GMIs, seroconversion rates and seropositive rates of the neutralizing antibody to SARS-CoV-2 Omicron strain (BA.1, BA.2), Prototype strain and Delta strain, induced by a booster dose of COVID-19 vaccine (Omicron variant) or Prototype COVID-19 vaccine, 28 days (Day 28) after booster vaccination among subjects with two-dose Prototype COVID-19 vaccine ≥6 months before
GMTs, GMIs, seroconversion rates and seropositive rates of the neutralizing antibody to SARS-CoV-2 Prototype strain (CZ strain) and Delta strain | 28 days (Day 28) after booster vaccination
  GMTs, GMIs, seroconversion rates and seropositive rates of the neutralizing antibody to SARS-CoV-2 Prototype strain (CZ strain) and Delta strain, induced by a booster dose of COVID-19 vaccine (Omicron variant) or Prototype COVID-19 vaccine, 28 days (Day 28) after booster vaccination among subjects with three-dose Prototype COVID-19 vaccine ≥6 months before
GMTs and seropositive rates of the neutralizing antibody to SARS-CoV-2 Prototype strain (CZ strain), Delta strain and Omicron strain (BA.1, BA.2) | 28 days after primary vaccination
  GMTs and seropositive rates of the neutralizing antibody to SARS-CoV-2 Prototype strain (CZ strain), Delta strain and Omicron strain (BA.1, BA.2), induced by two primary doses of Prototype COVID-19 vaccine in previous clinical trial serums, 28 days after primary vaccination
GMTs and seropositive rates of the neutralizing antibody to SARS-CoV-2 Omicron strain (BA.1, BA.2), Prototype strain (CZ strain) and Delta strain | 3 months (Day 90) and 6 months (Day 180) after booster vaccination
  GMTs and seropositive rates of the neutralizing antibody to SARS-CoV-2 Omicron strain (BA.1, BA.2), Prototype strain (CZ strain) and Delta strain, induced by one booster dose of COVID-19 vaccine (Omicron variant) or Prototype COVID-19 vaccine, 3 months (Day 90) and 6 months (Day 180) after booster vaccination among subjects with 2 or 3 doses of Prototype COVID-19 vaccine ≥6 months before
Incidence of local and systemic adverse reactions | within 0~7 days after booster vaccination
  Incidence of local and systemic adverse reactions within 0~7 days after booster vaccination among subjects with 2 or 3 doses of Prototype COVID-19 vaccine (CZ strain)
Incidence of serious adverse events (SAE) and adverse events of special interest (AESI) | 12 months after booster vaccination
  Incidence of serious adverse events (SAE) and adverse events of special interest (AESI) within 12 months after booster vaccination among subjects with 2 or 3 doses of Prototype COVID-19 vaccine (CZ strain)
Incidence of adverse reactions within 0~28 days | Within 0~28 days after booster vaccination
  Incidence of adverse reactions within 0~28 days after booster vaccination among subjects with 2 or 3 doses of Prototype COVID-19 vaccine (CZ strain)

OTHER OUTCOMES:
GMTs, GMIs, seroconversion rates and seropositive rates of the neutralizing antibody to SARS-CoV-2 Omicron strain (BA.1, BA.2), Prototype strain (CZ strain) and Delta strain | 7 days (Day 7) and 14 days (Day 14) after booster vaccination
  GMTs, GMIs, seroconversion rates and seropositive rates of the neutralizing antibody to SARS-CoV-2 Omicron strain (BA.1, BA.2), Prototype strain and Delta strain, induced by a booster dose of COVID-19 vaccine (Omicron variant) or Prototype COVID-19 vaccine (CZ strain), 7 days (Day 7) and 14 days (Day 14) after booster vaccination among subjects with two- or three-dose Prototype COVID-19 vaccine(CZ strain) ≥6 months before

CONTACTS AND LOCATIONS:
Overall Officials: Hongxing Pan, Master, Principal Investigator — Jiangsu Provincial Center for Disease Prevention and Control
Locations (1):
- Huaiyin Center for Disease Control and Prevention, Huai'an, Jiangsu, China

REFERENCES:
- [Background] Hu J, Liu Y, Liu S, Shu Q, Yang X, Chu K, Qiao Y, Hu Y, Wang K, Pan H. Safety and immunogenicity of a modified Omicron-adapted inactivated vaccine in healthy adults: a randomized, double-blind, active-controlled Phase III clinical trial. Front Immunol. 2023 Sep 18;14:1241153. doi: 10.3389/fimmu.2023.1241153. eCollection 2023. PMID 37799724